CLINICAL TRIAL: NCT05943444
Title: Comparison of Postoperative Anal Function Between Different Anastomosis Techniques(Parks Versus Bacon) in Low Rectal Cancer: A Prospective, Multicentric and Randomized Controlled Study
Brief Title: Comparison of Postoperative Anal Function Between Parks and Bacon Techniques in Low Rectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E2023072
Record Dates: First submitted 2023-06-28; First posted 2023-07-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Rectal Neoplasms; Low Anterior Resection Syndrome; Anastomotic Leak; Quality of Life
Keywords: anal function; Parks technique; Bacon technique
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome; Anastomotic Leak

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parks technique (Active Comparator): patients receive coloanal anastomosis operation
  Interventions: Procedure: Parks technique
- Bacon technique (Experimental): patients receive coloanal pull-out anastomosis operation
  Interventions: Procedure: Bacon technique

INTERVENTIONS:
Procedure: Parks technique — compare different operational styles of low rectal cancer
  Arms: Parks technique
Procedure: Bacon technique — Bacon technique
  Arms: Bacon technique

SUMMARY:
The goal of this study is to compare the postoperative anal function of patients with ultra-low rectal cancer after Parks operation (colon anal anastomosis) and Bacon operation (colon anal pull-out anastomosis), which may provide clinical evidence for the improvement of anal function and quality of life.

The main questions it aims to answer are: the difference of anal function 1 year after surgery type of study: clinical trial participant population: patients with low rectal cancer Participants will receive Parks operation of Bacon operation If there is a comparison group: Researchers will compare Parks and Bacon operation to see if the anal function 1 year after surgery is different.

DETAILED DESCRIPTION:
objective: To compare the postoperative anal function of patients with ultra-low rectal cancer after Parks operation (colon anal anastomosis) and Bacon operation (colon anal pull-out anastomosis), which may provide clinical evidence for the improvement of anal function and quality of life.

primary outcome: Low Anterior Resection Syndrome (LARS) score 1 year after surgery secondary outcomes: 1. LARS score at 3 months after surgery 2. LARS score at 6 months after surgery 3. Postoperative Quality of Life Score 4. The incidence of postoperative anastomotic complications

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, aged between 18 and 75 years;
2. Pathological diagnosis of rectal cancer before operation, with the distance from the lower edge of the tumor to the dentate line ≤ 3cm by MR imaging;
3. No local complications (including complete/ incomplete obstruction, active bleeding, local invasion of sphincter or levator ani, etc.) before operation;
4. Suitable for anal preservation surgery discussed by MDT;
5. Adequate bone marrow, liver, renal and cardiac function meeting the requirements of surgery and anesthesia;
6. R0 resection is expected technically;
7. Provision of written informed consent.

Exclusion Criteria:

1. Previous history of malignant colorectal tumors;
2. Complications such as obstruction and gastrointestinal bleeding that need an emergency operation;
3. Unachievable R0 resection due to invasion of adjacent organs by primary tumor;
4. Multiple primary tumors;
5. History of other malignancy;
6. Participation in other clinical trials within the previous 4 weeks of enrollment;
7. ASA physical status score ≥ IV level and/or ECOG performance status ≥ 2;
8. Intolerance of surgery due to liver, renal, cardiopulmonary or coagulation dysfunction, or underlying diseases;
9. History of serious mental disorders;
10. Women in pregnancy or lactation period;
11. Uncontrolled infection before operation;
12. Unsuitable to be included due to other clinical and laboratory conditions by the judgement of investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2027-08-08 (Estimated); Study Completion 2027-08-08 (Estimated)

PRIMARY OUTCOMES:
Low Anterior Resection Syndrome (LARS) score 1 year after surgery | 1 year after surgery
  use a scoring system for bowel dysfunction after LAR for rectal cancer on the basis of symptoms and impact on quality of life

SECONDARY OUTCOMES:
LARS score at 3 months after surgery | 3 months after surgery
  to score bowel dysfunction after LAR
LARS score at 6 months after surgery | 6 months after surgery
  to score bowel dysfunction after LAR
Postoperative Quality of Life Score | 3, 6, and 12 months after operation
  using a score system to access the quality of life after surgery
The incidence of postoperative anastomotic complications | 3, 6, and 12 months after operation
  the corresponding complications after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jun Huang, MD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital, Sun Yatsen University, Guangzhou, Guangdong, China